CLINICAL TRIAL: NCT05623930
Title: Hepatic Enzymes and Metabolic-Risk Factors Responses to Laser Acupuncture Versus Cupping Therapy in Fatty Liver
Brief Title: Liver Enzymes and Metabolic Risk Factors Response to Laser Acupuncture Versus Cupping Therapy in Fatty Liver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004116
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser on acupuncture points (Active Comparator): In fatty liver diseased patients which their number will be 30 patients, a 3-session/week application of 2-minute laser (for 3 months) on acupoint number 25,40,36 of stomach meridian, acupoints number 3 and 14 of liver meridian, acupoint number 6 of spleen meridian,acupoint number 9.12,4 of conception vessel meridian, acupoint number 14 of governor vessel meridian, acupoint number 4, 11 of large intestine meridian, acupoint number 34 of gall bladder meridian
  Interventions: Device: laser acupuncture
- cupping (with scarification) (Active Comparator): in this fatty liver diseased patients which their number will be 30, cupping (with scarification) or wet cupping will be applied at the first day and the day number 14 in the month for three successive months. cupping (with scarification) or wet cupping will be applied on urinary bladder acupoint 17 (on the both sides) and governosal vessels acupoints 12,13,and 14.
  Interventions: Other: wet cupping

INTERVENTIONS:
Device: laser acupuncture — In fatty liver diseased patients which their number will be 30 patients, a 3-session/week application of 2-minute laser (for 3 months) on acupoint number 25,40,36 of stomach meridian, acupoints number 3 and 14 of liver meridian, acupoint number 6 of spleen meridian,acupoint number 9.12,4 of conception vessel meridian, acupoint number 14 of governor vessel meridian, acupoint number 4, 11 of large intestine meridian, acupoint number 34 of gall bladder meridian
  Arms: laser on acupuncture points
Other: wet cupping — in this fatty liver diseased patients which their number will be 30, cupping (with scarification) or wet cupping will be applied at the first day and the day number 14 in the month for three successive months. cupping (with scarification) or wet cupping will be applied on urinary bladder acupoint 17 (on the both sides) and governosal vessels acupoints 12,13,and 14.
  Arms: cupping (with scarification)

SUMMARY:
fatty liver disease is characterized by low antioxidants, disturbed lipid metabolism, cardioautonomic functions, and elevated blood measures (glucose, inflammatory markers, liver enzymes)

DETAILED DESCRIPTION:
In fatty liver patients,applied cupping (with scarification) will be compared, regarding its effect on antioxidant, lipid metabolism, cardioautonomic functions, and blood measures (glucose, inflammatory markers, liver enzymes), to application of laser on acupoints

ELIGIBILITY:
Inclusion Criteria:

* fatty liver obese patients

Exclusion Criteria:

thoracic diseases heart diseases kidney diseases

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
high density lipoprotein | 12 weeks
  it is a component of lipid profile

SECONDARY OUTCOMES:
cholesterol | 12 weeks
  it is a component of lipid profile
low density lipoprotein | 12 weeks
  it is a component of lipid profile
triglycerides | 12 weeks
  it is a component of lipid profile
blood glucose | 12 weeks
  fasting level of blood glucose will be measured
C reactive protein | 12 weeks
  high sensitivity levels C reactive protein will be measured
Malondialdehyde | 12 weeks
  it ts oxidative stress marker
aspartate transaminase | 12 weeks
  it is a hepatic enzyme that reports the functions of liver
alanine transaminase | 12 weeks
  it is a hepatic enzyme that reports the functions of liver
systolic blood pressure | 12 weeks
  it will be measured by sphygmomanometer
diastolic blood pressure | 12 weeks
  it will be measured by sphygmomanometer
pulse rate | 12 weeks
  it will be measured manually

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt